CLINICAL TRIAL: NCT00616811
Title: A Multi-center, Randomized, Double-blind, Active-controlled Clinical Trial to Evaluate the Safety and Tolerability of 24 Weeks Treatment With Vildagliptin (50 mg qd) Versus Sitagliptin (25 mg qd) in Patients With Type 2 Diabetes and Severe Renal Insufficiency
Brief Title: Safety and Tolerability of Vildagliptin Versus Sitagliptin in Patients With Type 2 Diabetes and Severe Renal Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23138
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes, vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: vildagliptin
  Arms: Vildagliptin
Drug: Sitagliptin
  Arms: Sitagliptin

SUMMARY:
This clinical trial is designed to provide additional information on the safety and tolerability of vildagliptin (50 mg once daily (qd)) and sitagliptin (25 mg qd) when used in patients with type 2 diabetes mellitus(T2DM) and severe renal insufficiency (Glomerular filtration rate (GFR) < 30 mL/min) for a period of 24 weeks.

ELIGIBILITY:
Inclusion criteria

* History T2 DM
* Severe Renal Impairment

Exclusion criteria

* Glucose ≥ 270 mg/dL (≥15 mmol/L)
* Patients undergoing any method of dialysis
* Treatment with therapy other than sulfonylureas, TZDs ,insulin, and metiglinides

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in patients with T2DM and severe renal insufficiency over 24 weeks of treatment | 24 weeks

SECONDARY OUTCOMES:
Relationship between renal function and concentration levels of vildagliptin and its metabolites after repeated doses of vildagliptin in patients with T2DM and severe renal insufficiency. | 24 weekd
Efficacy of vildagliptin versus sitagliptin in patients with T2DM and severe renal insufficiency by assessing the hemoglobin A1c (HbA1c ) and fasting plasma glucose (FPG) reduction from baseline | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals
Locations (78):
- United States (78):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Anasazi Internal Medicine, Phoenix, Arizona
  - University of Arkanasas for Medical Sciences, Little Rock, Arkansas
  - Office of William Zigrang, Burlingame, California
  - John Muir Clinical Research, Concord, California
  - Academic Medical Research Institute, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Northern California Institute for Bone Health, Oakland, California
  - Dr. Wei Feng, Pasadena, California
  - Sierra Clinical Research - Orangevale, Roseville, California
  - Denver Nephrology PC, Denver, Colorado
  - Western Nephrology & Metabolic Bone Disease PC, Lakewood, Colorado
  - Western Nephrology & Metabolic Bone Disease PC, Westminster, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Nephrology Associates of South Miami, Aventura, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Center for Diabetes & Endocrine Care, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Osler Medical Clinical Research, Melbourne, Florida
  - Tampa Bay Nephrology Associates, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Boise Kidney & Hypertension Institiute, Meridian, Idaho
  - Iowa Diabetes & Endocrinology Research Center PLC, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - Cray Diabetes Education Center, Kansas City, Kansas
  - Cotton-O'Neil Diabetes & Endocrinology Center, Topeka, Kansas
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Metabolic Center of Louisiana, Baton Rouge, Louisiana
  - Bruce Samuels LLC, Covington, Louisiana
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Egan Healthcare, Metairie, Louisiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Northwest Louisiana Nephrology Research, Shreveport, Louisiana
  - Joslin Diabetes Center at North Arundel Hospital, Glen Burnie, Maryland
  - Biolab Research, LLC, Rockville, Maryland
  - Genesys Integrated Group Practice, PC, Flint, Michigan
  - Phillips Medical Services, PLLC, Jackson, Mississippi
  - Mississippi Medical Research, LLC, Picayune, Mississippi
  - Diabetes and Endocrinology Specialist, Inc, Chesterfield, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Arms, Dodge, Robinson, Wilber & Crouch, Inc., Kansas City, Missouri
  - Washington U School of Medicine, St Louis, Missouri
  - Platte Valley Medical Group, Kearney, Nebraska
  - Creighton Diabetes Center, Omaha, Nebraska
  - Creighton Nephrology, Omaha, Nebraska
  - UMDNJ-Robert Wood Johnson, New Brunswick, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Downstate University of Brooklyn, Brooklyn, New York
  - HRRG, Orchard Park, New York
  - Mayo Clinic Rochester, Rochester, New York
  - SUNY - Upstate Medical University, Syracuse, New York
  - Meritcare Medical Group, Fargo, North Dakota
  - Hightop Medical Research Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Lehigh Valley Hospital-Dept. of Medicine Research, Allentown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Renal Endocrine Associates, P. C., Pittsburgh, Pennsylvania
  - Aiken Center for Clinical Research, Aiken, South Carolina
  - Medical U of South Carolina, Charleston, South Carolina
  - SC Nephrology and Hyptertension Center, Inc., Orangeburg, South Carolina
  - Sumter Medical Specialists, Sumter, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Medical Nephrology Associates, Dyersburg, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Texas Tech University Health Sciences, El Paso, Texas
  - Baylor Clinic (BCM 621), Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Allied Institute of Medicine, San Antonio, Texas
  - Central Utah Clinic, American Fork, Utah
  - Clinical Research and Consulting Center, LLC, Fairfax, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - Washington State University at Spokane, Spokane, Washington
  - UW Health - West, Madison, Wisconsin

REFERENCES:
- [Derived] Kothny W, Lukashevich V, Foley JE, Rendell MS, Schweizer A. Comparison of vildagliptin and sitagliptin in patients with type 2 diabetes and severe renal impairment: a randomised clinical trial. Diabetologia. 2015 Sep;58(9):2020-6. doi: 10.1007/s00125-015-3655-z. Epub 2015 Jun 12. PMID 26067186
- See also: Results for CLAF237A23138 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4599